CLINICAL TRIAL: NCT04587323
Title: COVID-19 RELATED SUBMISSION: VEGF and sFlt-1 Levels in the Pathogenesis and Severity of COVID-19 Disease
Brief Title: VEGF and sFlt-1 Levels in the Pathogenesis and Severity of COVID-19 Disease
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Dylan R. Addis, MD, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300005378; UAB (Other: Anesthesiology)
Record Dates: First submitted 2020-09-22; First posted 2020-10-14 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: COVID-19 Disease
Keywords: COVID-19; SARS-CoV-2 viral infection; VEGF and sFlt-1 levels
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will identify patients with COVID-19 disease within the CCTS Biorepository with a blood (plasma) sample from within 7-14 days of symptom onset
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group 1:: Group 1: COVID-19 + inpatients who did not require mechanical ventilation (25 patients);
- Group 2:: Group 2: COVID-19 + inpatients who required mechanical ventilation (25 patients).
- Group 3:: Group 3: COVID-19 + inpatients with no preexisting cardiovascular disease (25 patients)
- Group 4:: Group 4: COVID-19 + inpatients with preexisting cardiovascular disease (25 patients).

SUMMARY:
To assess blood levels of vasoactive mediators that may regulate pulmonary endothelial permeability and contribute to multi-organ injury in patients with COVID-19 disease and to correlate the levels of these mediators with disease outcomes such as ICU admission, length of ventilatory support, respiratory failure, kidney failure, heart failure, and death.

DETAILED DESCRIPTION:
When patients are sick with other lung infections (pneumonias) caused by viruses or bacteria there are changes in a pathway that regulates the "leakiness" the tiny airspaces inside the lungs. Even bigger changes in this pathway are seen when patients develop severe breathing difficulties (acute respiratory distress syndrome) similar to what is seen in patients who get really sick with COVID-19 disease.

There are important changes in this pathway that occur in patients who have preexisting cardiovascular (heart) disease who do not have lung infections. The investigator will evaluate these levels in patients with COVID-19 because the investigator believes that this baseline difference in pathway regulation may be one reason patients with heart disease who contract COVID-19 get sicker than patients without heart or vascular disease.

The investigator will also assess the levels of components of this pathway in patients who are less sick with those who became sick enough to require a tube to help them breathe because this is important to determine if COVID-19 lung disease has a similar effect on this pathway as other lung infections like flu and bacterial pneumonias.

ELIGIBILITY:
Inclusion Criteria:

* Positive test for COVID-19 (SARS-CoV-2 infection)
* >=18 years
* Blood (plasma) specimen(s) available in the CCTS biorepository

Exclusion Criteria:

* <18 years
* Lack of blood specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have available specimens in the UAB CCTS Biorepository for COVID-19 patients. (IRB-300005127: COVID-19 Enterprise Biorepository.)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-22 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Laboratory Assays | 7-14 days after symptom onset
  The primary outcome measure is the ratio of soluble fms-like tyrosine kinase receptor-1 (sFlt-1) to vascular endothelial growth factor (VEGF) which will be obtained using an immunoassay on blood samples. The specimens will be analyzed using enzyme-linked immunosorbent assay and reported as a ratio
VEGF-A | 7-14 days after symptom onset
  Plasma samples will be analyzed to measure VEGF-A
VEGF-C | 7-14 days after symptom onset
  Plasma samples will be analyzed to measure VEGF-C
VEGF-D | 7-14 days after symptom onset
  Plasma samples will be analyzed to measure VEGF-D
Tie-2 | 7-14 days after symptom onset
  Plasma samples will be analyzed to measure Tie-2
Flt-1 | 7-14 days after symptom onset
  Plasma samples will be analyzed to measure Flt-1
PlGF | 7-14 days after symptom onset
  Plasma samples will be analyzed to measure PlGF
FGF | 7-14 days after symptom onset
  Plasma samples will be analyzed to measure FGF

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Addis, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States